CLINICAL TRIAL: NCT03476694
Title: Effects of Various Volume of Local Anaesthetic Use for Ultrasound Guided Supraclavicular Brachial Plexus Block on Successful Blockade and Diaphragmatic Motility.
Brief Title: Ultrasound Guided Supraclavicular Brachial Plexus Block, Volume Comparison of Local Anaesthetics and Diaphragmatic Motility.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Shambhu Adhikari, Resident doctor, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRC/1091/017
Record Dates: First submitted 2018-03-18; First posted 2018-03-26 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Sucessful Block With Less Hemidiaphragmatic Paresis in Distal Upper Arm Fracture

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 20ml of 0.75% Ropivacine (Experimental)
  Interventions: Procedure: ultra sound guided supraclavicular brachial plexus block
- 25ml of 0.75% Ropivacine (Experimental)
  Interventions: Procedure: ultra sound guided supraclavicular brachial plexus block

INTERVENTIONS:
Procedure: ultra sound guided supraclavicular brachial plexus block — ultra sound guided supraclavicular brachial plexus block , comparing the volume of 0.75 % ropivacine in sucessful block and hemidiaphragmatic motilty.

SUMMARY:
Brachial plexus block as done by landmark technique use large volume of local anaesthetics (at least 30-40 ml), leading to higher incidence of phrenic nerve involvement and diaphragmatic dysfunction. With use of ultrasound dose of local anaesthetic can be reduced. Volume as low as 20 ml when use by ultrasound guidance has shown to provide successful block with no hemidiaphragmatic palsy when compared with nerve stimulation technique. But no study has compared the different volumes of drug on success rate and diaphragmatic motility.So in this study , the investigators want to compare the incidence of hemidiaphragm paralysis and success of block with different volumes of local anaesthetic , so that the lowest effective dose with higher safety profile can be determined.

ELIGIBILITY:
Inclusion

* Age between 18 and 60 years undergoing distal arm surgery
* American Society of Anesthesiologists physical status 1 to 3
* Able to give informed consent
* Body weight greater than 50 kg

Exclusion

* Patient refusal for supraclavicular block.
* Inability to obtain informed consent.
* Contraindication to Brachial plexus block
* Pulmonary and cardiac disorders
* Pregnancy
* Allergy to local anesthetic
* Chest or shoulder deformities

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
hemidiaphragmatic paralysis | within 30 minutes after sucessfull blocade
  grading of hemidiaphragmatic paralysis as, complete ,partial and no hemidiaphragmatic paralysis as reduction of diaphragmatic excursion greater than 75%, 25-75%, less than 25% respectively after sucessful blocade.

SECONDARY OUTCOMES:
sucessful blocade | within 30 minutes of block
  ultrasound guided supraclavicular brachial plexus block using ropivacine and observing the complete block.

CONTACTS AND LOCATIONS:
Locations (1):
- B P Koirala Institute of Health science (BPKIHS), Dharān, Koshi Zone, Nepal

IPD SHARING:
Plan to Share IPD: No